CLINICAL TRIAL: NCT02536924
Title: Randomized Control Trial of RESOLVE (Relaxation Exercise, SOLving Problem and cognitiVe Errors): A Waiting Room Intervention for Crisis Clients
Brief Title: RCT of RESOLVE: A Waiting Room Intervention for Crisis Clients
Acronym: RESOLVE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Queen's University (Other)
Responsible Party: Principal Investigator, Dr. Farooq Naeem, Principal Investigator, Queen's University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 6015290
Record Dates: First submitted 2015-08-29; First posted 2015-09-01 (Estimated); Last update posted 2015-09-01 (Estimated); Status verified 2015-08

CONDITIONS: Depression Anxiety Disorder
MeSH Terms: interventions — Therapeutics

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Waiting room intervention plus TAU (Experimental): The treatment group will receive waiting room intervention plus treatment as usual.
  Interventions: Behavioral: Waiting Room Intervention; Behavioral: Treatment as usual.
- Only TAU. (Experimental): The control group will receive only treatment as usual.
  Interventions: Behavioral: Treatment as usual.

INTERVENTIONS:
Behavioral: Waiting Room Intervention — The waiting room intervention is called RESOLVE (Relaxation SOLving problem and cognitive errors), which is a short film.
  Arms: Waiting room intervention plus TAU
Behavioral: Treatment as usual. — The patient will receive treatment as usual.

SUMMARY:
Crisis Teams are now a well established part of the mental health system. These teams are effective in providing crisis management, treatment, referral, and educational services. We are testing a waiting room intervention for the patients attending a Crisis Team. As far as we are aware, no trial of a waiting room intervention has been reported in a psychiatric setting. This is a preliminary study using a Randomized Control Trial (RCT) Design. Patients (N =40) will be randomly allocated to either the treatment or the control group, and will be selected from the local Crisis Team. The treatment group will receive a waiting room intervention called, RESOLVE (Relaxation, SOLving problem and cognitiVe Errors), that is a short film, Plus Treatment As Usual (TAU), and the control group will receive only TAU. Patients in both groups will be assessed before and after the intervention, using the HADS (Hospital Anxiety And Depression Scale), CORE (Clinical Outcome in Routine Evaluation), (to measure psychopathology) and WHODAS (World Health Organization Disability Assessment Schedule) (for functioning). We hypothesize that the treatment group will demonstrate significant improvement in mental health and functioning, compared to the control group. Analyses will be conducted using SPSS v22, and will consist of a t-test or Chi Square test to measure the baseline differences, and a linear regression to compare the differences between the two groups at the end of the intervention. Results will be published in international journals and will be presented in local and international conferences.

DETAILED DESCRIPTION:
GRANT APPLICATION The mental health crisis teams are now a well established and vital part of the mental health system. These teams are uniquely equipped to provide front-line mental health care when and where it is most needed. It is able to provide on-site assessment, crisis management, treatment, referral, and educational services to patients, families, law enforcement officers, and the community at large. Mental health crisis teams provide access to mental health care for even the most under-served populations efficiently and cost-effectively. The cost-effectiveness of the team's services is defined by savings in both monetary and human terms (Zealberg, Santos, & Fisher, 1993) (Scott, 2000). However, no interventions have been developed, that are specific to this service.

Patients attending the crisis teams usually wait for their appointments, just like other health settings. This can be a valuable time that can be used to deliver short term educational interventions. This has been tried and tested in general health settings (Coyne, Palmer, Shapiro, Thompson, & DeMichele, 2004; Holmes-Garrett, 1990; Oermann, n.d.; Rhodes et al., 2001; Wheeler et al., 2001). As far as we are aware no waiting room interventions have been tried or tested in psychiatric setup. We have developed an intervention RESOLVE (Relaxation Exercise, SOLving problem and cognitiVe Errors), that can be easily delivered using eMedia (for example a tv screen) in waiting room. This intervention is short enough to be given while patients are in a waiting room in a psychiatric clinic. A crisis team setting might be ideal as most patients might find a problem solving approach helpful. We want to conduct a pilot using a Randomised Controlled Trial design (RCT) to assess effectiveness of this intervention.

METHODS Objectives The primary objective of this preliminary pilot study is to assess the effectiveness of a "waiting room intervention" for patients attending a crisis clinic. The objectives of the study are to see if the intervention can reduce (1) symptoms of depression and anxiety, (2) overall psychopathology, and (3) disability.

Participants Participants (N =40) will be primarily recruited from the Crisis Clinic in Kingston. Inclusion criteria are; All those who fulfill the diagnostic criteria of Depressive episode (F32) or Recurrent depressive disorder (F33 except 33.4 ) using ICD10 RDC, are between the ages of 18 to 65. Patients will be asked to attend a further appointment at the end of study period and will be assessed again. The exclusion criteria include; excessive use of alcohol or drugs (using ICD 10 RDC for alcohol or drug abuse or dependence) significant cognitive impairment (for example learning disability or dementia) and active psychosis. Data will be kept strictly confidential, available only to the primary investigators. Participants may withdraw from the study at any time without penalties.

Study design This preliminary evaluation will use a Randomized Control Trial (RCT) design. Randomization will be performed using www.randomization.com, from the list of all the patients who consent. Study participants will be randomly assigned to either treatment or the control arm. The treatment group will receive waiting room intervention plus TAU (Treatment As Usual), while the control group will receive only TAU. Patients who have been referred for the study will be provided brief information about the study. Those who meet the criteria and consent will be then asked to join the study and will be allocated to one arm of the trial after randomization.

Measurements Demographic information will be collected using a short questionnaire. Assessments will be carried out by two research assistants independently. We will also collect data on number of contacts with the Crisis Team, number of admissions and duration of contact with the Crisis Team.

The Hospital Anxiety and Depression Scale (HADS) (Zigmond and Snaith, 1983) is a 14 item, self assessment scale designed to measure anxiety and depression. It has a high internal consistency, face validity and concurrent validity. Even-numbered questions relate to depression and odd-numbered questions relate to anxiety. Each question has 4 possible responses. Responses are scored on a scale from 3 to 0. The maximum score is therefore 21 for depression and 21 for anxiety. A score of 11 or higher indicates the probable presence of the mood disorder with a score of 8 to 10 being just suggestive of the presence of the respective state. The two subscales, anxiety and depression, have been found to be independent measures. In its current form the HADS is now divided into four ranges: normal (0-7), mild (8-10), moderate (11-15) and severe (16-21).

The Clinical Outcome in Routine Evaluatoin (CORE) is is a client self-report questionnaire designed to be administered before and after therapy. The client is asked to respond to 34 questions about how they have been feeling over the last week, using a 5-point scale ranging from 'not at all' to 'most or all of the time'. The 34 items of the measure cover four dimensions: Subjective well-being, Problems/symptoms, Life functioning and Risk/harm. The responses are designed to be averaged by the practitioner to produce a mean score to indicate the level of current psychological global distress (from 'healthy' to 'severe'). The questionnaire is repeated after the last session of treatment; comparison of the pre-and post-therapy scores offers a measure of 'outcome' (i.e. whether or not the client's level of distress has changed, and by how much) (Evans, 2000).

The World Health Organization Disability Assessment Schedule 2.0 (WHODAS) (Ustün et al., 2010) will be used to measure functioning. This scale assesses disability due to physical and psychological problems, and has been used extensively in research settings.

Procedure Patients who fulfill the inclusion criteria will be provided with information about the study. Those who consent in writing will be randomly allocated to one arm of the trial. All participants will complete the demographics questionnaire, HADS, WHO DAS & CORE during an interview with a primary investigator. Participants in the treatment arm will attend 1 session of the intervention in addition to the Treatment As Usual. Participants in the control group will receive treatment as usual during this time. Participants in both groups will be assessed at the end of 3 months wand then 6 months post intervention.

Data entry and analysis Statistical analyses will be carried out using an Intention To Treat, using SPSS v22. Both parametric and non-parametric tests will be carried out as appropriate to compare groups. Treatment and control groups will be compared at the baseline, using Chi square and t test. A linear regression will be used to compare the two groups at the end of assessment period. This will be done, using group as the independent, and the end of assessment scores as dependent variables. Baseline scores and variables that are not equally distributed in two groups will be used as covariates. All the analyses will be carried out by FN.

Results and Research Implications If effective, this innovative intervention will reduce distress, psychopathology and disability in this group and will possibly improve functioning. Success with this preliminary study could lead to subsequent research to further investigate this novel intervention.

Description of Research Team

1. Tariq Munshi: Primary Investigator- will co-supervise and train the team and will help with recruitment
2. Farooq Naeem: Co-Investigator- will supervise Research Assistants as they conduct the study; will conduct statistical analyses 3 Neeraj Bajjaj- Co-Investigator- will co-supervise the team and will help with recruitment

ELIGIBILITY:
Inclusion Criteria:

* All those who fulfill the diagnostic criteria of Depressive episode (F32) or Recurrent depressive disorder (F33 except 33.4) using ICD10 RDC
* between the ages of 18-65
* must meet the assessment criteria at the beginning and the end of the study period

Exclusion Criteria:

* excessive use of alcohol or drugs (using ICD 10 RDC for alcohol or drug abuse or dependence)
* significant cognitive impairment (for example learning disability or dementia)
* active psychosis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2015-08; Primary Completion 2016-08 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
Hospital Anxiety and Depression Scale (HADS) | 6 months
  14 item, self assessment scale designed to measure anxiety and depression.

SECONDARY OUTCOMES:
The Clinical Outcome in Routine Evaluation (CORE) | 6 months
  A client self-report questionnaire designed to be administered before and after therapy.
World Health Organization Disability Assessment Schedule 2.0 (WHODAS) | 6 months
  A client self-report questionnaire designed to be administered before and after therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Farooq Naeem, MSc, PhD, Principal Investigator — Queen's University
Locations (1):
- Addiction & Mental Health Services- Kingston Frontenac Lennox and Addington, Kingston, Ontario, Canada

REFERENCES:
- [Background] Coyne JC, Palmer SC, Shapiro PJ, Thompson R, DeMichele A. Distress, psychiatric morbidity, and prescriptions for psychotropic medication in a breast cancer waiting room sample. Gen Hosp Psychiatry. 2004 Mar-Apr;26(2):121-8. doi: 10.1016/j.genhosppsych.2003.08.012. PMID 15038929
- [Background] Evans, J. M.-C., Frank Margison, Michael Barkham, Kerry Audin, Janice Connell, Graeme McGrath, Chris. (2000). CORE: Clinical Outcomes in Routine Evaluation. Journal of Mental Health, 9(3), 247-255. http://doi.org/10.1080/jmh.9.3.247.255
- [Background] Holmes-Garrett, C. (1990). The Crisis of the Forgotten Family. Social Work with Groups, 12(4), 141-157. http://doi.org/10.1300/J009v12n04_09
- [Background] Oermann MH. Effects of educational intervention in waiting room on patient satisfaction. J Ambul Care Manage. 2003 Apr-Jun;26(2):150-8. doi: 10.1097/00004479-200304000-00007. PMID 12698929
- [Background] Rhodes KV, Lauderdale DS, Stocking CB, Howes DS, Roizen MF, Levinson W. Better health while you wait: a controlled trial of a computer-based intervention for screening and health promotion in the emergency department. Ann Emerg Med. 2001 Mar;37(3):284-91. doi: 10.1067/mem.2001.110818. PMID 11223765
- [Background] Scott RL. Evaluation of a mobile crisis program: effectiveness, efficiency, and consumer satisfaction. Psychiatr Serv. 2000 Sep;51(9):1153-6. doi: 10.1176/appi.ps.51.9.1153. PMID 10970919
- [Background] Wheeler JG, Fair M, Simpson PM, Rowlands LA, Aitken ME, Jacobs RF. Impact of a waiting room videotape message on parent attitudes toward pediatric antibiotic use. Pediatrics. 2001 Sep;108(3):591-6. doi: 10.1542/peds.108.3.591. PMID 11533323
- [Background] Zealberg JJ, Santos AB, Fisher RK. Benefits of mobile crisis programs. Hosp Community Psychiatry. 1993 Jan;44(1):16-7. doi: 10.1176/ps.44.1.16. No abstract available. PMID 8436356
- [Derived] Naeem F, Munshi T, Gratzer D, Rodie D, Irfan M, Rao S, Husain N, Farooq S, Sanches M, Ayub M, Lecomte T. Video intervention for the psychiatric waiting room: proof-of-concept randomised controlled trial of RESOLVE (Relaxation Exercise, SOLVing problem and cognitive Errors). BJPsych Open. 2019 Sep 6;5(5):e77. doi: 10.1192/bjo.2019.59. PMID 31488227